CLINICAL TRIAL: NCT02741895
Title: Using Wearable Biosensors to Monitor Ambulation After Major Surgery: Optimizing Efficiency of Postoperative Recovery
Brief Title: Using Fitbit to Monitor Ambulation in Patients After Surgery.
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Timothy J. Daskivich, Assistant Professor, Urology Academic Practice, Cedars-Sinai Medical Center
Other Study IDs: Pro00044059
Record Dates: First submitted 2016-04-12; First posted 2016-04-18 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: General Surgery
Keywords: Biosensing Techniques; Patient Readmission

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Postoperative patients: The target populations for the study are patients undergoing robotic cystectomy, open colectomy, abdominal hysterectomy, esophagectomy, lung lobectomy, gastric bypass, and hip replacement at Cedars-Sinai Medical Center.
  Interventions: Behavioral: Fitbit monitoring

INTERVENTIONS:
Behavioral: Fitbit monitoring — Patients will be fitted with a Fitbit after surgery, which will monitor steps and active minutes for the duration of hospitalization.

SUMMARY:
This study will evaluate whether information on postoperative ambulation from Fitbits can improve surgeons' ability to monitor ambulation and identify patients at risk for prolonged length of stay, 30-day readmissions, and discharge to transitional care after major surgery.

DETAILED DESCRIPTION:
After the patient is awake and alert after surgery, a study team member will place the Fitbit device on participants' wrists. Investigators will then monitor daily steps taken and active minutes for the duration of hospitalization, with the option to discontinue if clinically required or requested by the patient or provider. Investigators will record the wearable biosensor number and subject study number on a secure spreadsheet.

To supplement Fitbit data, a research coordinator will collect clinical data from chart review of the electronic health record (age, gender, race/ethnicity, body mass index, comorbid health conditions), and enter the data into a secure spreadsheet.

Physicians will also be participating in the study by providing data on estimated daily ambulation, using a standard formatted scale. Surgeons currently assess daily ambulation in the medical record, but assessments are not uniform, which precludes meaningful comparisons between providers. Investigators will therefore ask physicians to record daily estimates of ambulatory status according to standardized terms that are commonly used in the medical record (nonambulatory; out of bed to chair; out of bed to ambulate (QD, BID, TID); and ambulating ad lib). Investigators will also collect information on daily ambulation orders as entered by the provider team as part of routine practice. This information will be ascertained by chart review and entered into the secure spreadsheet along with the additional patient data.

The Fitbit device has a battery life of approximately 7 days, so investigators will plan to recharge and download information every 5 days.

At the time of discharge, a study team member will remove the device and download the information from the device to a secure spreadsheet. The wearable biosensor will be reset at that time and the information will be erased from its memory. Investigators will also clean the wearable biosensors with disinfectant used for durable medical equipment.

Investigators will also query the medical record for information regarding disposition outcomes, including length of stay (from end of surgery to discharge from the hospital) and location of disposition (to home, rehab facility, or skilled nursing facility). Investigators will then contact the patients by phone after 30 days have elapsed since discharge to inquire whether they have been readmitted to the hospital or ER within the 30 days of their discharge date.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Undergoing robotic cystectomy, open colectomy, abdominal hysterectomy, esophagectomy, lung lobectomy, gastric bypass, or hip replacement
* Able to provide informed consent

Exclusion Criteria:

1. Unable to provide consent
2. Not undergoing procedure of interest
3. Admitted to ICU directly after operation (except esophagectomy, where all patients are admitted to ICU directly after the operation)
4. Use of walker, cancer, or wheelchair at baseline
5. Presence of physical limitations on walking (i.e. amputation)
6. Usual place of residence is skilled nursing facility
7. Cognitive inability to follow directions to maintain biosensor in place
8. Unable to place biosensor on patient's wrist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical inpatients who have undergone one of the following: robotic cystectomy, open colectomy, abdominal hysterectomy, esophagectomy, lung lobectomy, gastric bypass, or hip replacement.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Location of disposition | Through study completion, on average 1 week
  Home, Rehab Facility, or Skilled Nursing Facility
30-day readmission | 30 days post discharge
  Presence or absence of readmission to hospital or ER visit within 30 days of discharge.
Number of steps | Through study completion, on average 1 week
  Number of steps per day during hospitalization, per Fitbit data.
Active minutes | Through study completion, on average 1 week
  Active minutes per day during hospitalization, per Fitbit data.
Physician daily assessment of ambulatory status | Through study completion, on average 1 week
  Physician daily assessment of ambulatory status
Length of stay | Through study completion, on average 1 week
  Days from admission (end time of surgery) until discharge from hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Daskivich, MD, MSHPM, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
We have not yet considered a plan to share data.

REFERENCES:
- [Background] Chandrasekaran S, Ariaretnam SK, Tsung J, Dickison D. Early mobilization after total knee replacement reduces the incidence of deep venous thrombosis. ANZ J Surg. 2009 Jul;79(7-8):526-9. doi: 10.1111/j.1445-2197.2009.04982.x. PMID 19694660
- [Background] Garcia Guerrero JJ, Fernandez de la Concha Castaneda J, Lopez Quero D, Collado Bueno G, Infante de la Torre JR, Rayo Madrid JI, Redondo Mendez A. Lower incidence of venous thrombosis with temporary active-fixation lead implantation in mobile patients. Europace. 2010 Nov;12(11):1604-7. doi: 10.1093/europace/euq262. Epub 2010 Jul 28. PMID 20667893
- [Background] Pearse EO, Caldwell BF, Lockwood RJ, Hollard J. Early mobilisation after conventional knee replacement may reduce the risk of postoperative venous thromboembolism. J Bone Joint Surg Br. 2007 Mar;89(3):316-22. doi: 10.1302/0301-620X.89B3.18196. PMID 17356141
- [Background] Kamel HK, Iqbal MA, Mogallapu R, Maas D, Hoffmann RG. Time to ambulation after hip fracture surgery: relation to hospitalization outcomes. J Gerontol A Biol Sci Med Sci. 2003 Nov;58(11):1042-5. doi: 10.1093/gerona/58.11.m1042. PMID 14630887
- [Background] Delaney CP, Zutshi M, Senagore AJ, Remzi FH, Hammel J, Fazio VW. Prospective, randomized, controlled trial between a pathway of controlled rehabilitation with early ambulation and diet and traditional postoperative care after laparotomy and intestinal resection. Dis Colon Rectum. 2003 Jul;46(7):851-9. doi: 10.1007/s10350-004-6672-4. PMID 12847356
- [Background] Rath S, Schreuders TA, Stam HJ, Hovius SE, Selles RW. Early active motion versus immobilization after tendon transfer for foot drop deformity: a randomized clinical trial. Clin Orthop Relat Res. 2010 Sep;468(9):2477-84. doi: 10.1007/s11999-010-1342-4. Epub 2010 Apr 17. PMID 20401554
- [Background] Browning L, Denehy L, Scholes RL. The quantity of early upright mobilisation performed following upper abdominal surgery is low: an observational study. Aust J Physiother. 2007;53(1):47-52. doi: 10.1016/s0004-9514(07)70061-2. PMID 17326738
- [Background] Larsen K, Hansen TB, Thomsen PB, Christiansen T, Soballe K. Cost-effectiveness of accelerated perioperative care and rehabilitation after total hip and knee arthroplasty. J Bone Joint Surg Am. 2009 Apr;91(4):761-72. doi: 10.2106/JBJS.G.01472. PMID 19339559
- [Background] Kalisch BJ, Landstrom GL, Hinshaw AS. Missed nursing care: a concept analysis. J Adv Nurs. 2009 Jul;65(7):1509-17. doi: 10.1111/j.1365-2648.2009.05027.x. Epub 2009 May 9. PMID 19456994
- [Background] Kalisch BJ, Tschannen D, Lee H, Friese CR. Hospital variation in missed nursing care. Am J Med Qual. 2011 Jul-Aug;26(4):291-9. doi: 10.1177/1062860610395929. Epub 2011 Jun 3. PMID 21642601
- [Background] Brown CJ, Friedkin RJ, Inouye SK. Prevalence and outcomes of low mobility in hospitalized older patients. J Am Geriatr Soc. 2004 Aug;52(8):1263-70. doi: 10.1111/j.1532-5415.2004.52354.x. PMID 15271112
- [Background] Callen BL, Mahoney JE, Grieves CB, Wells TJ, Enloe M. Frequency of hallway ambulation by hospitalized older adults on medical units of an academic hospital. Geriatr Nurs. 2004 Jul-Aug;25(4):212-7. doi: 10.1016/j.gerinurse.2004.06.016. PMID 15311196
- [Background] Collins FS, Varmus H. A new initiative on precision medicine. N Engl J Med. 2015 Feb 26;372(9):793-5. doi: 10.1056/NEJMp1500523. Epub 2015 Jan 30. PMID 25635347
- [Background] Topol EJ. The creative destruction of medicine : how the digital revolution will create better health care. 1st pbk. ed. New York: Basic Books; 2013.
- [Background] Augustyniak P. Wearable wireless heart rate monitor for continuous long-term variability studies. J Electrocardiol. 2011 Mar-Apr;44(2):195-200. doi: 10.1016/j.jelectrocard.2010.11.014. PMID 21353066
- [Background] Shambroom JR, Fabregas SE, Johnstone J. Validation of an automated wireless system to monitor sleep in healthy adults. J Sleep Res. 2012 Apr;21(2):221-30. doi: 10.1111/j.1365-2869.2011.00944.x. Epub 2011 Aug 22. PMID 21859438
- [Background] Spiegel BM, Kaneshiro M, Russell MM, Lin A, Patel A, Tashjian VC, Zegarski V, Singh D, Cohen SE, Reid MW, Whitman CB, Talley J, Martinez BM, Kaiser W. Validation of an acoustic gastrointestinal surveillance biosensor for postoperative ileus. J Gastrointest Surg. 2014 Oct;18(10):1795-803. doi: 10.1007/s11605-014-2597-y. Epub 2014 Aug 5. PMID 25091837
- [Background] Appelboom G, Yang AH, Christophe BR, Bruce EM, Slomian J, Bruyere O, Bruce SS, Zacharia BE, Reginster JY, Connolly ES Jr. The promise of wearable activity sensors to define patient recovery. J Clin Neurosci. 2014 Jul;21(7):1089-93. doi: 10.1016/j.jocn.2013.12.003. Epub 2013 Dec 9. PMID 24534628
- [Background] Dobkin BH. Wearable motion sensors to continuously measure real-world physical activities. Curr Opin Neurol. 2013 Dec;26(6):602-8. doi: 10.1097/WCO.0000000000000026. PMID 24136126
- [Background] Dobkin BH, Dorsch A. The promise of mHealth: daily activity monitoring and outcome assessments by wearable sensors. Neurorehabil Neural Repair. 2011 Nov-Dec;25(9):788-98. doi: 10.1177/1545968311425908. PMID 21989632
- [Background] Kalisch BJ, Lee S, Dabney BW. Outcomes of inpatient mobilization: a literature review. J Clin Nurs. 2014 Jun;23(11-12):1486-501. doi: 10.1111/jocn.12315. Epub 2013 Sep 13. PMID 24028657
- [Background] ATKINSON GS. Early post-operative ambulation. Clin Med (Northfield). 1948 Dec;55(12):245. No abstract available. PMID 18107881